CLINICAL TRIAL: NCT06967220
Title: The Impact of Inflammation on Skeletal Muscle Maintenance in Hospitalized Patients
Acronym: InflaMus
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Grith Højfeldt, Principle Investigator, Bispebjerg Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: BBH170
Record Dates: First submitted 2025-04-17; First posted 2025-05-13 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-04

CONDITIONS: Disease Related Malnutrition; High Systemic Inflammation; Geriatric Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anti-inflammatory diet and supplements (Experimental): A sub group of patients with high inflammation will be offered a diet where 50% of the regular hospital diet is switched for diet containing plant based food and nutrients found to lower inflammation
  Interventions: Other: Single leg training

INTERVENTIONS:
Other: Single leg training — All subjects will train one leg twice daily.

SUMMARY:
The main goal is to elucidate the mechanistic coupling between inflammation and the ability to maintain skeletal muscle through physical exercise while hospitalized. We will investigate protein kinetics in patients who belong to one of three groups 1) high inflammatory state, 2) moderate inflammatory state and 3) low/no inflammation. We will further intervene in group 1 (high inflammatory state) with anti-inflammatory nutrition (primarily green-solution plant-based) to diminish activity in inflammatory pathways. The hypothesis is that inflammation will inhibit protein synthesis in skeletal muscle both in resting muscle and in strength trained skeletal musculature, and that a lowering of the inflammatory status by anti-inflammatory nutrition will enhance the exercise induced formation of new muscle mass. .

ELIGIBILITY:
Inclusion Criteria:

* Hospitalised at the geriatric department at Bispebjerg Hospital with an expected admission time of minimum 7 days
* Have Disease Related Malnutrition (DRM)
* Able to carry out strength training
* Able to understand the study information, as assessed by the research team

Exclusion Criteria:

* Current use of anti-inflammatory medication
* Liver failure
* Short bowel syndrome
* Chrohn's or colitis
* Terminally ill

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2026-04-22 (Estimated); Study Completion 2026-04-22 (Estimated)

PRIMARY OUTCOMES:
FSR in high vs. low inflammation group | 7 days (or until hospital discharge)
  The primary outcome is the muscle protein fractional synthesis rate (FSR) in the high inflammation group vs. the low inflammation group

SECONDARY OUTCOMES:
Change in muscle size between groups | 7 days (or until hospital discharge)
  Change in muscle size during the study period between the three groups
FSR in trained vs. non trained leg | 7 days (or until hospital discharge)
  Effect of training on the muscle protein fractional synthesis rate
Inflammation in regular vs. antiinflammatory diet | 7 days (or until hospital discharge)
  Comparison of the changes in plasma C-Reactive Protein (CRP) from day 1 till discharge between the group ingesting regular diet vs. the group ingesting an anti-inflammatory diet.
AA uptake following feeding | 7 days (or until hospital discharge)
  Plasma amino acid profile following a standard meal
Muscle size in trained vs. untrained leg | 7 days (or until hospital discharge)
  The difference in muscle size in trained vs. untrained leg measured using ultrasound
Change in muscle strength between groups | 7 days (or until discharge)
  Description: Change in muscle strength during the study period between the three groups. Hand muscle strength is measured using a hand dynamometer, and leg muscle strength (MVC) is measured using an isokinetic dynamometer.
  Time Frame: 7 days (or until hospital discharge)
Muscle strength in trained vs. untrained leg | 7 days (or until hospital discharge)
  The difference in leg muscle strength (MVC) in trained vs. untrained leg measured using an isokinetic dynamometer.

OTHER OUTCOMES:
Feasibility of training | 7 days (or until hospital discharge)
  It will be reported if the subjects can complete a minium of 80% of the twice-daily training sessions.

CONTACTS AND LOCATIONS:
Locations (1):
- Bispebjerg Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided